CLINICAL TRIAL: NCT04670367
Title: Baduanjin Exercise on Cardiac Surgery
Brief Title: The Effects of Baduanjin Exercise on Meridian Energy and Heart Rate Variability in Patients Undergoing Cardiac Sugery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Chun Hou Huang, Assistance Professor, Tzu Chi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: TCU-CHHuang-BaduanjinHeart
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Open Heart Surgery
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: usual care (Placebo Comparator): routine usual care
  Interventions: Other: usual care
- Arm B: walk (Experimental): walk 30mins per day, 5 days per week.
  Interventions: Behavioral: Walk 30mins
- Arm C: Baduanjin (Experimental): Baduanjin 12 mins per day, 5 days per week.
  Interventions: Behavioral: Baduanjin
- Arm D: Baduanjin plus walk (Experimental): walk 30mins then Baduanjin 12 mins per day, 5 days per week.
  Interventions: Behavioral: Walk plus Baduanjin

INTERVENTIONS:
Behavioral: Walk 30mins — aerobic exercise
  Arms: Arm B: walk
Behavioral: Walk plus Baduanjin — Walk 30mins then Baduanjin 12mins per day, 5 times per week.
  Arms: Arm D: Baduanjin plus walk
Other: usual care — routine care
  Arms: Arm A: usual care
Behavioral: Baduanjin — Baduanjin exercise is moderate in intensity and short in duration (a set of Baduanjin takes about 12 minutes). Baduanjin consists of the sitting and standing practicing form. The sitting Baduanjin exercise conforms to the aspects of low-intensity and long-term aerobic activity, which is suitable for the rehabilitation training of patients who are in stable condition during hospitalization. The standing Baduanjin is more suitable for patients with sequential rehabilitation after discharge and can be adjusted based on the patient's condition
  Arms: Arm C: Baduanjin

SUMMARY:
Cardiac rehabilitation (CR) consists of supervised exercise training in conjunction with other secondary prevention interventions. However, CR is not widely used because of distance, financial resources, work and other time constraints, gender, age, social support, illness perceptions, and psychiatric problems. Baduanjin is a type of movement-based mind-body intervention. It is a form of traditional practice designed to promote physical and psychological health, manage symptoms, and relieve stress during illness. Patients with heart disease have frequently used it. The impacts of a Baduanjin exercise-based cardiac rehabilitation program for patients recovering from CAD under coronary artery bypass graft (CABG) or valve replacement on Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) and heart rate variability (HRV) has yet to be assessed. This trial evaluates whether the Baduanjin exercise would provide effective meridian energy and HRV in patients following CABG.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 age range
* Undergoing open heart surgery
* Hemodynamically stable
* Ambulatory
* No advanced vision defect
* The physician authorized by the operating physician for participation in the exercise
* Patients who agreed to participate in the study.

Exclusion Criteria:

* The presence of pulmonary, neurological, musculoskeletal disease limiting participation in exercise training
* Patients at high risk (ejection fraction below 40 percent)
* Dissectant aneurysm
* Patients who cannot be cooperative in verbal and / or auditory terms
* Psychological and / or perceptual cooperative patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-05-27 (Estimated); Study Completion 2022-11-27 (Estimated)

PRIMARY OUTCOMES:
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing open-heart surgery as assessed using M.E.A.D (Meridian Energy Analysis Device)：Baseline | Baseline
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current.Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing open-heart surgery as assessed using M.E.A.D (Meridian Energy Analysis Device)： 2 weeks | 2 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current.Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing open-heart surgery as assessed using M.E.A.D (Meridian Energy Analysis Device)： 4 weeks | 4 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current.Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing open-heart surgery as assessed using M.E.A.D (Meridian Energy Analysis Device)： 12 weeks | 12 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current.Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing open-heart surgery as assessed using M.E.A.D (Meridian Energy Analysis Device)： 16 weeks | 16 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current.Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No